CLINICAL TRIAL: NCT07306351
Title: The Effect of Recovery Training on Lower Extremity Explosive Strength in Tennis Players
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, alyildirim, PhD, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1669
Record Dates: First submitted 2025-11-25; First posted 2025-12-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy Tennis Players
Keywords: Recovery training; Explosive strength; Tennis player; Sports performance

STUDY DESIGN:
Intervention Model Description: The experimental group will receive recovery training in addition to routine tennis training.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants in this group will continue their regular tennis training
- Recovery Training Group (Experimental): Participants in this group will continue their regular tennis training and additionally perform recovery training twice a week for four weeks. The recovery sessions include stretching, foam rolling, and relaxation exercises designed to enhance recovery and improve lower extremity explosive strength.
  Interventions: Other: Recovery Training Group

INTERVENTIONS:
Other: Recovery Training Group — Participants in this group will continue their regular tennis training and additionally perform recovery training twice a week for four weeks. The recovery sessions include stretching, foam rolling, and relaxation exercises designed to enhance recovery and improve lower extremity explosive strength.
  Arms: Recovery Training Group

SUMMARY:
This study was designed to examine the effects of recovery training on lower extremity explosive strength performance in tennis players. Recovery methods are known to play an important role in reducing muscle fatigue, accelerating the recovery process, and decreasing the risk of injury among athletes. However, the effects of recovery training on lower extremity explosive strength in tennis players have not been sufficiently investigated in the literature.

This study will be conducted as a randomized controlled experimental design. Volunteer athletes aged 11-17 who regularly play tennis will be included in the study. Participants will be randomly divided into two groups: the control group will continue only their regular tennis training, while the experimental group will receive additional recovery training along with their routine tennis sessions. Lower extremity explosive strength will be evaluated using the countermovement jump, squat jump, reactive strength index (RSI), standing long jump, single-leg hop, and single-leg vertical jump tests. Measurements will be performed before and after the six-week training period.

The findings obtained from this research will scientifically reveal the contribution of recovery training to performance improvement in tennis players and provide evidence-based insights for optimizing athlete health and training program design.

ELIGIBILITY:
Inclusion Criteria:

* Must be 11-18 years old and have been playing tennis for the past year.
* Must be cooperative.
* Must have participated in regular tennis training for at least 2 years.
* Must have no history of acute lower extremity injury before the study.
* Must be voluntary and have signed an informed consent form from the athlete and/or their parent.

Exclusion Criteria:

* Having a history of acute injury, fracture, surgery, or chronic musculoskeletal problems affecting the lower extremity
* Having a neurological or cardiovascular disease
* Having taken a break from sports due to a serious lower extremity injury within the last 6 months

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Countermovement Jump Height | 4 weeks
  The countermovement jump (CMJ) test was used to assess lower extremity explosive performance. Participants started from an upright standing position with hands placed on the hips. Following a rapid downward movement involving hip and knee flexion, participants immediately performed a maximal vertical jump. Jump height (cm) was recorded using [measurement device - e.g., force plate / jump mat / Optojump system]. The CMJ reflects the efficiency of the stretch-shortening cycle and is considered a reliable indicator of explosive lower limb performance.
Squat Jump Height | 4 weeks
  The squat jump (SJ) test was used to assess concentric lower extremity explosive performance. Participants started from a semi-squat position with approximately 90° of hip and knee flexion, with hands placed on the hips. After holding this position briefly to eliminate the contribution of elastic energy, participants performed a maximal vertical jump without a preparatory countermovement. Jump height (cm) was recorded using [measurement device - e.g., force plate / jump mat / Optojump system]. The SJ test allows direct evaluation of concentric muscle power of the lower limbs.
Reactive Strength Index | 4weeks
  RSI is a performance measure that reflects reactive strength and neuromuscular efficiency. It is typically assessed through a drop jump in which the participant steps off a platform, lands, and performs a quick rebound jump with minimal ground contact time. RSI is sensitive to the athlete's ability to rapidly switch from eccentric to concentric action, a capacity highly relevant to sports requiring explosive changes in direction, such as tennis .
Standing Long Jump | 4 weeks
  SLJ, also known as the broad jump, is a field-based test for assessing horizontal explosive strength of the lower extremities. The participant stands with feet shoulder-width apart, swings the arms, and jumps forward as far as possible. The landing distance, measured from the starting line to the heel mark, reflects the ability of the lower-limb muscles to generate forward propulsion .
Single-Leg Hop for Distance | 4 weeks
  SLH test evaluates unilateral lower-limb performance and limb symmetry. The participant stands on one leg, performs a maximal forward hop, and lands on the same leg while maintaining balance for at least two seconds. Distances are recorded for both legs, and comparisons provide valuable insights into side-to-side asymmetries, rehabilitation status, and injury risk.
Single-Leg Vertical Jump Height | 4 weeks
  The single-leg vertical jump (SLVJ) test was used to assess unilateral lower extremity explosive performance. Participants stood on one leg with hands placed on the hips, while the non-supporting leg was flexed and held stationary. From a stable standing position, participants performed a maximal vertical jump using the supporting leg only. Jump height (cm) was recorded separately for each limb using [measurement device - e.g., force plate / jump mat / Optojump system]. This test allows evaluation of unilateral vertical force production and identification of inter-limb asymmetries.is .

CONTACTS AND LOCATIONS:
Locations (1):
- Sportplus Tennis Academy, Istanbul, Maltepe, Turkey (Türkiye)

REFERENCES:
- [Result] Markovic G, Mikulic P. Neuro-musculoskeletal and performance adaptations to lower-extremity plyometric training. Sports Med. 2010 Oct 1;40(10):859-95. doi: 10.2165/11318370-000000000-00000. PMID 20836583
- [Result] Moran J, Ramirez-Campillo R, Granacher U. Effects of Jumping Exercise on Muscular Power in Older Adults: A Meta-Analysis. Sports Med. 2018 Dec;48(12):2843-2857. doi: 10.1007/s40279-018-1002-5. PMID 30341594
- [Result] Ebben WP, Petushek EJ. Using the reactive strength index modified to evaluate plyometric performance. J Strength Cond Res. 2010 Aug;24(8):1983-7. doi: 10.1519/JSC.0b013e3181e72466. PMID 20634740
- [Result] Castro-Pinero J, Ortega FB, Artero EG, Girela-Rejon MJ, Mora J, Sjostrom M, Ruiz JR. Assessing muscular strength in youth: usefulness of standing long jump as a general index of muscular fitness. J Strength Cond Res. 2010 Jul;24(7):1810-7. doi: 10.1519/JSC.0b013e3181ddb03d. PMID 20555277
- [Result] Gustavsson A, Neeter C, Thomee P, Silbernagel KG, Augustsson J, Thomee R, Karlsson J. A test battery for evaluating hop performance in patients with an ACL injury and patients who have undergone ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2006 Aug;14(8):778-88. doi: 10.1007/s00167-006-0045-6. Epub 2006 Mar 9. PMID 16525796
- [Result] Meylan C, McMaster T, Cronin J, Mohammad NI, Rogers C, Deklerk M. Single-leg lateral, horizontal, and vertical jump assessment: reliability, interrelationships, and ability to predict sprint and change-of-direction performance. J Strength Cond Res. 2009 Jul;23(4):1140-7. doi: 10.1519/JSC.0b013e318190f9c2. PMID 19528866
- [Result] Dupuy O, Douzi W, Theurot D, Bosquet L, Dugue B. An Evidence-Based Approach for Choosing Post-exercise Recovery Techniques to Reduce Markers of Muscle Damage, Soreness, Fatigue, and Inflammation: A Systematic Review With Meta-Analysis. Front Physiol. 2018 Apr 26;9:403. doi: 10.3389/fphys.2018.00403. eCollection 2018. PMID 29755363